CLINICAL TRIAL: NCT04424693
Title: A Prospective Randomized Clinical Research Trial Comparing the Incidence of Preeclampsia Between Pregnant Women Receiving Tdap Vaccinations at Week 28 and Those Receiving Tdap Vaccinations at Week 36
Brief Title: Comparing the Incidence of Preeclampsia Between Pregnant Women Receiving Tdap Vaccinations at Week 28 or at Week 36
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Arthritis Research (Other)
Collaborators: Louisiana State University Health Sciences Center in New Orleans (Other); Brigham Young University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PE-Tdap01
Record Dates: First submitted 2020-06-03; First posted 2020-06-11 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Pre-Eclampsia; Diphtheria, Tetanus and Pertussis Vaccine Reaction
Keywords: Preeclampsia; Tdap vaccinations
MeSH Terms: conditions — Pre-Eclampsia; Diphtheria; Tetanus

STUDY DESIGN:
Intervention Model Description: Pregnant women enlisted in the double blinded study will be randomized to receive Tdap vaccination either at week 28 or week 36 and observed and treated with standard of care.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each study site will designate an "injection nurse" who will be responsible for preparing both placebo and Tdap administration and will be the only one knowing when a patient gets either Tdap injection at week 28 or placebo injection at week 28, or gets Tdap injection at week 36 or placebo injection at week 36. This person will be the only one at each site who will know the randomization of each subject and is the only one who will administer the injection. Every subject will receive Tdap either at week 28 or week 36 and receive placebo injection on the other injection time.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tdap vaccinations at gestational week 28 (Active Comparator): Pregnant women entering into this clinical research study and signing informed consent at week 12 will be randomized to either receive Tdap vaccination at week 28 or week 36. Subjects receiving Tdap vaccination at week 28 will receive a placebo injection at week 36. Subject will be followed with routine standard of care throughout their pregnancy and have routine clinic visits from which study visits will include weeks 12, 20, 28, 36, and 2 weeks postpartum. Data will be collected at each of these visits with special attention to the development of preeclampsia and fetal health
  Interventions: Drug: Tdap Vaccine Administration
- Tdap vaccinations at gestational week 36 (Active Comparator): Pregnant women entering into this clinical research study and signing informed consent at week 12 will be randomized to either receive Tdap vaccination at week 28 or week 36. Subjects receiving Tdap vaccination at week 36 will receive a placebo injection at week 28. Subjects will be followed with routine standard of care throughout their pregnancy and have routine clinic visits from which study visits will include weeks 12, 20, 28, 36, and 2 weeks postpartum. Data will be collected at each of these visits with special attention to the development of preeclampsia and fetal health
  Interventions: Drug: Tdap Vaccine Administration

INTERVENTIONS:
Drug: Tdap Vaccine Administration — Tdap vaccinations are routinely given during pregnancy between weeks 27 and 36 per guidelines of American College Obstetrics and Gynecology (ACOG) -- but this study uniquely is trying to establish that the earlier Tdap vaccinations reduce preeclampsia by more than 50%

SUMMARY:
Preeclampsia is a significant medical condition occurring in 3-8% of pregnancies and impacts deleteriously both maternal and fetal health. An important discovery has been made by Dr Craig D Scoville showing that early Tdap vaccinations in pregnancy can reduce the incidence of preeclampsia by more than 50%. A prospective clinical research trial is proposed and urgently needed to validate this finding and thereby make a significant contribution in reducing the incidence of this common and severe complication of pregnancy.

DETAILED DESCRIPTION:
A double blinded randomized prospective clinical research study is proposed to validate the hypothesis that Tdap vaccinations at week 28 in pregnancy can reduce the incidence of preeclampsia by more than 50%. This project will recruit 1600 pregnant women with appropriate informed consent in the first trimester of pregnancy, obtain detailed obstetric and health history, and then randomize these subjects so 800 women receive Tdap at week 28, and 800 women receive Tdap at week 36, and all women will be followed during their pregnancies using standard of care with special attention to preeclampsia and fetal outcomes. Blood samples will be obtained at weeks 12, 20, and 36 in order to test the anti-tetanus toxoid antibody levels, anti-diptheria antibody levels, anti-pertussis antibody levels, and also maternal cytokines (IL-2, IL-4, IL-6, IL-10, TNFa, IL-17, and IFNg), and placental biomarkers (sFlt-1, sEng, and PIGF) for preeclampsia on those patients who develop preeclampsia and compare to those who didn't and thereby better understand the biomarkers of preeclampsia and devise a better formula for positive prediction for preeclampsia. To make this change in clinical practice and save lives, this study is asking for funding from NICHD PA-18-480.

ELIGIBILITY:
Inclusion Criteria:

1. confirmed pregnancy at week 12
2. Age 18 to 42
3. Willing to participate and sign informed consent documentation
4. willing to follow study procedures with regards to randomization of Tdap and attend all routine clinic visits per obstetrician and standard of care
5. accept Tdap vaccination either at week 28 or week 36

Exclusion Criteria:

1. no history of allergic reaction or intolerance to Tdap vaccination
2. No history of cancer in past 5 years prior to this study (except for non melanoma localized skin cancers or cancer in situ) -

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 1600 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of preeclampsia in each arm of the study with regards to timing of Tdap vaccination | Through duration of pregnancy approximately 10 months
  The definition of preeclampsia in this study will follow the guidelines of ACOG inclusive of hypertension, proteinuria, but also other features
Incidence of preeclampsia in each arm of the study with regards to the quantitative anti-tetanus toxoid antibody level | Through duration of pregnancy approximately 10 months
  Test the hypothesis that pregnant women with anti-tetanus toxoid antibody levels <1.0 IU/ml are at higher risk of preeclampsia compared to those with higher levels. Obtain blood levels for anti-tetanus toxoid antibody levels, anti-pertussis antibody levels, and anti-diptheria antibody levels will be tested at weeks 12, 20, and 36

SECONDARY OUTCOMES:
Assessment of other potential risk factors for preeclampsia inclusive of BMI, hypertension, prior history of preeclampsia, first pregnancy | Through duration of pregnancy approximately 10 months
  Statistical analysis of all possible variables for preeclampsia

OTHER OUTCOMES:
Compare the placental and maternal biomarkers of preeclampsia in order to devise a better formula for positive prediction of preeclampsia | Through duration of pregnancy at 12, 20 and 36 week of gestation
  Follow the quantitative levels of maternal cytokines in pg/ml: IL-2, IL-4, IL-6, IL-10, TNFa, IL-17, IFNg and placental biomarkers in pg/ml PIGF during pregnancy at weeks 12, 20, and 36 and compare these levels with those women who develop preeclampsia to normal pregnancy cohorts from this study during the same times tested
Compare the placental and maternal biomarkers of preeclampsia in order to devise a better formula for positive prediction of preeclampsia | Through duration of pregnancy at 12, 20 and 36 week of gestation
  Follow the quantitative levels of maternal placental biomarkers in ng/ml sFlt-1 and sEng during pregnancy at weeks 12, 20, and 36 and compare these levels with those women who develop preeclampsia to normal pregnancy cohorts from this study during the same times tested

CONTACTS AND LOCATIONS:
Overall Officials: Craig D Scoville, MD, PhD, Principal Investigator — Institute of Arthritis Research
Locations (1):
- Institute of Arthritis Research, Idaho Falls, Idaho, United States

IPD SHARING:
Plan to Share IPD: Yes
Data acquired in this project will be shared through presentations at scientific meetings and published peer reviewed publications. In order to disseminate the data, we will maintain a data archive where all information is stored and can be distributed. Data requests may be sent to the PI and reasonable requests will be granted. However a particular data set in the archives will only be shared after a manuscript describing the main findings has been accepted for publication. Also any proprietary information will not be shared until legal restrictions make it permissible
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: see Plan Description and no time limit once the data is made available to the public
Access Criteria: contact Institute of Arthritis Research at scovilleclinic.com